CLINICAL TRIAL: NCT00583219
Title: Botulin-A Toxin/Dimethyl Sulfoxide Bladder Instillations for Treatment of Voiding Dysfunction Secondary to Detrusor Hyperreflexia and Detrusor Instability in Women
Brief Title: Botulin-A Toxin Instillations and Overactive Bladder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr. Steven Petrou, Mayo Clinic Jacksonville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 359-06
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Overactive Bladder; Detrusor Instability; Detrusor Hyperreflexia
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; incobotulinumtoxinA; Dimethyl Sulfoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botox/DMSO Solution (Experimental): Subjects received Botulinum-A toxin and Dimethyl sulfoxide solution. The first 3 subjects in Phase 1 underwent bladder instillation of 50 cc of the solution utilizing 200 units of botulinum-A toxin and 50cc DMSO. The next 6 subjects in the Phase 1 trial received 300 units of botulinum-A toxin and 50cc DMSO.
  All subjects in the Phase 2 trial received 300 units of botulinum-A toxin and 50cc DMSO.
  Interventions: Drug: Botulinum-A toxin; Drug: Dimethyl sulfoxide (DMSO)

INTERVENTIONS:
Drug: Botulinum-A toxin — A simple bladder catheterization in the office with a standard urinary catheter and instill the Botulinum-A toxin/DMSO solution.
  Other Names: Botox; Dysport; Xeomin
Drug: Dimethyl sulfoxide (DMSO) — Subjects received 50 cc of DMSO in an aqueous solution for intravesical instillation with botulinum-A toxin. Each cc contained 0.54 gm DMSO.

SUMMARY:
The primary objective of this pilot study is to evaluate the safety and efficacy of direct instillations of Botulinum-A toxin/DMSO into the bladder via a catheter system as a means of treating women with symptoms of overactive bladder and secondary urinary incontinence. In doing so, we will focus on estimating the percentage of women who experience an improvement in their urinary incontinence symptoms at one month and three months following this novel instillation technique.

DETAILED DESCRIPTION:
Rationale:

To date, the standard treatment for overactive bladder (including detrusor hyperreflexia and detrusor overactivity) consists of oral anticholinergic medications that can have troublesome side effects and variable efficacy. What's more, patients failing pharmacological therapy must either live with their malady or undergo open surgery that is irreversible and carries a prolonged convalescence. The fact remains however that treatment for overactive bladder is necessary to help maintain quality of life and prevent upper urinary tract deterioration. In recent years, cystoscopic-guided injection of Botulinum-A toxin has been used as a novel method of addressing detrusor hyperreflexia and overactivity by blocking acetylcholine transmission at the bladder. The obvious benefits of a more targeted therapy notwithstanding, this method requires the use of a cystoscope, needle delivery of the agent through approximately 30 separate injection sites and either regional or topical intravesical anesthesia for peri-operative pain control. Clearly, the identification of less invasive and more cost effective means of delivering the beneficial effects of Botulinum-A toxin to the bladder muscle has the potential to enhance the overall appeal of this treatment method.

Objectives:

The primary objective of this pilot study is to evaluate the safety and efficacy of direct instillations of Botulinum-A toxin/DMSO into the bladder via a catheter system as a means of treating women with symptoms of overactive bladder and secondary urinary incontinence. In doing so, we will focus on estimating the percentage of women who experience an improvement in their urinary incontinence symptoms at one month and three months following this novel instillation technique.

Study Design:

We are proposing a single center, Phase II pilot study for this investigation. In this proposal, 25 sterile women between 18-90 years of age with urodynamic evidence of detrusor overactivity, hyperreflexia or symptoms of overactive bladder syndrome who lack evidence of infection and stress incontinence will be offered bladder instillation of Botulinum-A toxin with DMSO as a carrier agent if they have failed anticholinergic medications or cannot tolerate the pharmacological side effects. We will use two validated measurement tools for determining urinary incontinence severity. These measurement tools will be administered to each women at baseline and then again at one month and three-month follow-up time points. Our analysis will also focus on identifying and describing adverse events among these women and estimating the percentage of women that experience a successful improvement in their urinary incontinence symptoms.

Study Duration:

Patients will sign an informed consent and be screened for eligibility. Once determined eligible for the study, each patient will be scheduled for baseline evaluation and instillation of Botox/DMSO. Patients will be then followed up at one month and three months. Patients will be removed from the study if they withdraw consent, experience one of the study stopping criteria (in which case the entire study will stop) or when they complete the final follow-up evaluation at three-months.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient aged 18 years or older
2. Patient with a history of stress urinary incontinence for at least 12 months
3. Patient with Intrinsic Sphincter Deficiency who demonstrate an abdominal leak point pressure of less than 100 cm of water on urodynamic evaluation
4. Patient with urinary incontinence verified by the Provocation test: a mean urinary leakage of 10 g on screening and baseline visits
5. Patient with positive stress test and/or urodynamic stress incontinence
6. Patient who has failed prior non-invasive treatment (e.g. behavior modification, pelvic floor exercises, biofeedback, electrical stimulation and/or drug therapy)
7. Patient with negative Contigen skin test during screening.
8. Patient who is mentally competent with the ability to understand and comply with the requirements of the study
9. Patient who agrees to be available for the follow-up evaluations as required by the protocol
10. Patient who has given signed informed consent

Exclusion Criteria:

1. Patient with Q-tip angle greater than 30 degrees
2. Patient with Functional Bladder capacity <200 ml as recorded in the baseline Bladder Diary
3. Patient with Post-Void Residual Urine (PVRU) greater than 100 ml on repeated measures. (Patient with a single PVRU of >100 ml and followed by two consecutive PVRU measurements of <100 ml may be included in the study)
4. Patient with vesicoureteral reflux, interstitial cystitis, genitourinary fistulae
5. Patient with predominant urge incontinence
6. Patient with detrusor overactivity on filling cystometry
7. Patient with pelvic organ prolapse stage III or IV, i.e. the most distal part of the prolapse protruding more than 1 cm beyond the hymen (>+1), at straining
8. Patient with urinary incontinence due to neurological disease that is known to affect urinary tract infection
9. Patient with uninvestigated hematuria
10. Patient with genitourinary malignancies
11. Patient on current medication for stress urinary incontinence, such as alpha-adrenergic agonists or duloxetine, within three weeks prior to completing the baseline Bladder Diary (estrogen therapy on a stable dose for at least two months prior to study start is allowed)
12. Patient who has had bulking therapy for stress urinary incontinence
13. Patient with ongoing complications of prior anti-incontinence surgery
14. Patient who is pregnant, lactating, or planning to become pregnant within the study period
15. Patient who has received pelvic radiation
16. Patient with any condition, which could lead to significant postoperative complications, including current infection and uncontrolled diabetes.
17. Patient who is morbidly obese (defined as BMI > 32 Kg/m2)
18. Patient who is bedridden, institutionalized or in such physical condition that she cannot move to the closest bathroom without assistance from another person
19. Patient with current or acute urinary tract infection, including cystitis or urethritis. (Patient with such infections should be treated with antibiotics, with subsequent urinalysis tests confirming the absence of such infection before study inclusion)
20. Patient with any condition that would preclude treatment due to contraindications and/or warnings in the study product's labeling
21. Patient on concomitant medication with anticoagulant properties (e.g., Warfarin, Heparin, Aspirin, Nonsteroidal anti-inflammatory drugs (NSAIDs), except for cox-2 inhibitors) within two weeks prior to treatment
22. Patient on immunomodulatory therapy (suppressive or stimulatory)
23. Patient with a known allergy to bovine collagen
24. Patient with known lidocaine hypersensitivity or hypersensitivity to any anesthetics to be used during the treatment session/surgical procedure
25. Patient with a concurrent use of another study product within two weeks prior to study start, or who concurrently participate in any other clinical study
26. Any disease that in the opinion of the Investigator would make the patient unsuitable for the study
27. Patient with a life expectancy of less than 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Petrou, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States

REFERENCES:
- [Result] Petrou SP, Parker AS, Crook JE, Rogers A, Metz-Kudashick D, Thiel DD. Botulinum a toxin/dimethyl sulfoxide bladder instillations for women with refractory idiopathic detrusor overactivity: a phase 1/2 study. Mayo Clin Proc. 2009 Aug;84(8):702-6. doi: 10.4065/84.8.702. PMID 19648387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from November 2006 to March 2009 at Mayo Clinic in Jacksonville, Florida.
Groups:
- Botox/DMSO Solution: Subjects received Botulinum-A toxin and Dimethyl sulfoxide solution. The first 3 subjects in Phase 1 underwent bladder instillation of 50 cc of the solution utilizing 200 units of botulinum-A toxin and 50cc DMSO. The next 6 subjects in the Phase 1 trial received 300 units of botulinum-A toxin and 50cc DMSO.
  All subjects in the Phase 2 trial received 300 units of botulinum-A toxin and 50cc DMSO.
  Botulinum-A toxin: A simple bladder catheterization in the office with a standard urinary catheter and instill the Botulinum-A toxin/DMSO solution.
  Dimethyl sulfoxide (DMSO): Subjects received 50 cc of DMSO in an aqueous solution for intravesical instillation with botulinum-A toxin. Each cc contained 0.54 gm DMSO.
Period: Phase 1
Arm/Group | Botox/DMSO Solution
Started | 9 (First 3 subjects in Phase 1 received 200 units Botox. The remaining subjects got 300 units Botox.)
Completed | 9
Not Completed | 0
Period: Phase 2
Arm/Group | Botox/DMSO Solution
Started | 22 (6 subjects from P1 continued in P2; plus 16 new subjects. All subjects in P2 got 300 units Botox.)
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Botox/DMSO Solution: Subjects received Botulinum-A toxin and Dimethyl sulfoxide solution. The first 3 subjects in Phase 1 underwent bladder instillation of 50 cc of the solution utilizing 200 units of botulinum-A toxin and 50cc DMSO. The next 6 subjects in the Phase 1 trial received 300 units of botulinum-A toxin and 50cc DMSO.
  The 6 subjects in the Phase 1 trial who received 300 units of botulinum-A toxin and 50cc DMSO also continued in the Phase 2 trial. All subjects in the Phase 2 trial received 300 units of botulinum-A toxin and 50cc DMSO.
  Botulinum-A toxin: A simple bladder catheterization in the office with a standard urinary catheter and instill the Botulinum-A toxin/DMSO solution.
  Dimethyl sulfoxide (DMSO): Subjects received 50 cc of DMSO in an aqueous solution for intravesical instillation with botulinum-A toxin. Each cc contained 0.54 gm DMSO.
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 74 [37 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Body Mass Index [Median (Full Range); unit: kg/m^2] | 26.6 [18.4 to 40.0]

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Incontinent Episodes During 24 Hours
Description: The study coordinator instructed the subject to keep record of any incontinence episodes during the 24-hour period prior to their baseline and follow-up visits.
Time Frame: baseline, 1 month, 3 months
Measure: Median (Inter-Quartile Range); unit: number of incontinent episodes
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
number of incontinent episodes
  Baseline | 4 [2 to 9]
  1 month | 2 [0 to 5]
  3 months | 4 [2 to 6]
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline at one month; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Botox/DMSO Solution; P value change from baseline to 3 months; Test type: Superiority or Other; p = 0.81, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Median 24 Hour Pad Weight
Description: Prior to baseline and follow-up visits, the study coordinator weighed standard pads provided to the subject for the study time period. The study coordinator instructed the subject to bring in any pads used during the 24-hour period prior to baseline and follow up visits. The study coordinator recorded the 24-hour pad weights into the study dataset.
Time Frame: baseline, 1 month, 3 months
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
g
  Baseline | 135 [6 to 259]
  1 month | 46 [9 to 183]
  3 months | 55 [11 to 318]
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline to 1 month; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Botox/DMSO Solution; P value change from baseline to 3 months; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Blaivas-Groutz Anti-Incontinence Score at Baseline
Description: The Blaivas-Groutz Anti-incontinence scale was used as a measure of urinary incontinence. This scale combines information on the number of incontinent episodes in a 24-hour period, 24-hour pad weights, and a qualitative rating by the patient into a single score ranging from 0 to 6. This score is then used to categorize incontinence as none (0), mild (1-2), moderate (3-4), or severe (5-6).
Time Frame: baseline
Measure: Number; unit: participants (per category)
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
participants (per category)
  None | 0
  Mild | 4
  Moderate | 1
  Severe | 16

4. Secondary Outcome: Blaivas-Groutz Anti-Incontinence Score at 1 Month
Description: as for outcome 3
Time Frame: 1 month after treatment
Measure: Number; unit: participants (per category)
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
participants (per category)
  None | 1
  Mild | 5
  Moderate | 5
  Severe | 10
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Blaivas-Groutz Anti-Incontinence Score at 3 Months
Description: as for outcome 3
Time Frame: 3 months after treatment
Measure: Number; unit: participants (per category)
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
participants (per category)
  None | 0
  Mild | 2
  Moderate | 6
  Severe | 13
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline; Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Mean Number of Pads Per Day
Time Frame: baseline, 1 month, 3 months
Measure: Mean (Inter-Quartile Range); unit: pads per day
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
pads per day
  Baseline | 4 [2 to 7]
  1 month | 3 [1 to 5]
  3 months | 3 [2 to 5]
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline to 1 month; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Botox/DMSO Solution; P value change from baseline to 3 months; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Postvoid Residual
Time Frame: baseline, 1 month, 3 months
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
mL
  Baseline | 8 [0 to 24]
  1 month | 19 [0 to 32]
  3 months | 24 [9 to 65]
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline to 1 month; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Botox/DMSO Solution; P value change from baseline to 3 months; Test type: Superiority or Other; p = 0.033, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Urine Culture
Time Frame: baseline, 1 month, 3 months
Measure: Number; unit: participants
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
participants
  baseline negative | 16
  baseline positive | 5
  1 month negative | 16
  1 month positive | 5
  3 months negative | 13
  3 months positive | 8
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline to 1 month; Test type: Superiority or Other; p > 0.99, Exact binomial sign test
Statistical Analysis 2: Comparison: Botox/DMSO Solution; P value change from baseline to 3 months; Test type: Superiority or Other; p = 0.25, exact binomial sign test

9. Secondary Outcome: Urinary Urgency at Baseline
Description: Urinary urgency was measured by the Indevus Urgency Severity Scale (IUSS). The IUSS asks patients to assess the severity of 'urgency' at each void. The scale employs the following wording: "Degree of urgency is meant to describe your urge to urinate. Sometimes you may feel a very strong urge to urinate and at other times, you may feel a milder urge prior to the onset of a toilet void. Rate this feeling by circling 0, 1, 2, or 3, defined as: 0: NONE - no urgency, 1: MILD - awareness of urgency, but it is easily tolerated and you can continue with your usual activity or tasks, 2: MODERATE - enough urgency discomfort that it interferes with or shortens your usual activity or tasks, 3: SEVERE - extreme urgency discomfort that abruptly stops all activity or tasks."
Time Frame: baseline
Measure: Number; unit: participants (per category)
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
participants (per category)
  None | 0
  Mild | 2
  Moderate | 8
  Severe | 11

10. Secondary Outcome: Urinary Urgency at 1 Month
Description: as for outcome 9
Time Frame: 1 month after treatment
Measure: Number; unit: participants (per category)
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
participants (per category)
  None | 0
  Mild | 13
  Moderate | 7
  Severe | 1
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline to one month; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Urinary Urgency at 3 Months
Description: as for outcome 9
Time Frame: 3 months after treatment
Measure: Number; unit: participants (per category)
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
participants (per category)
  None | 0
  Mild | 11
  Moderate | 7
  Severe | 3
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Median Urogenital Distress Inventory (UDI-6) Scores
Description: The UDI-6 was one measure of urinary-associated quality of life. The UDI-6 questionnaire has 6 items, scored from 0 (not at all) to 3 (greatly), with total scores ranging from 0 to 18, a higher score indicating greater distress.
Time Frame: baseline, 1 month, 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
units on a scale
  Baseline | 10 [8 to 12]
  1 month | 5 [4 to 9]
  3 months | 6 [4 to 8]
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline to 1 month; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Botox/DMSO Solution; P value change from baseline to 3 months; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Bothersomeness
Description: The bothersomeness refers to the question: On a scale of 1-10 (0 is not at all; 10 is intolerable), how badly does loss of urinary control bother you?
Time Frame: baseline, 1 month, 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
units on a scale
  Baseline | 9 [8 to 10]
  1 month | 5 [3 to 8]
  3 months | 5 [2 to 7]
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline to one month; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Botox/DMSO Solution; P value change from baseline to 3 months; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Incontinence Impact Questionnaire-short Form (IIQ-7) Scores
Description: The IIQ-7 was one measure of urinary-associated quality of life. The IIQ-7 questionnaire has 7 items, scored from 0 (not at all) to 3 (greatly), with total scores ranging from 0 to 21, a higher score indicating greater distress.
Time Frame: baseline, 1 month, 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Botox/DMSO Solution
Number analyzed (Participants) | 21
units on a scale
  Baseline | 13 [10 to 18]
  1 month | 7 [2 to 11]
  3 months | 6 [2 to 12]
Statistical Analysis 1: Comparison: Botox/DMSO Solution; P value change from baseline to 1 month; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Botox/DMSO Solution; P value change from baseline to 3 months; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Phase 1 patients (9) were assess immediately, 4 hours 24 hours, and 7 days after instillation. Phase 2 patients were assessed immediately, 2 hours, and 4 hours after instillation. All patients were assessed at 1 month and 3 month follow-up intervals.
Arm/Group | Botox/DMSO Solution
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 18/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox/DMSO Solution (N=25)
Pelvic soreness in first 24 hours (Renal and urinary disorders) | 1 (1)
Positional light-headedness in first 24 hours (General disorders) | 1 (1)
Anxiety in first 24 hours (Psychiatric disorders) | 1 (1)
Bladder spasms in first 24 hours (Renal and urinary disorders) | 2 (2)
Urethral discomfort in first 24 hours (Renal and urinary disorders) | 2 (2)
Dysuria in first 24 hours (Renal and urinary disorders) | 2 (2)
Urinary tract infection after 24 hours (Renal and urinary disorders) | 3 (3)
Perineal rash 7 days after injection (Reproductive system and breast disorders) | 1 (1)
Throbbing with urination 7 days after injection (Renal and urinary disorders) | 1 (1)
Dysuria after 24 hours (Renal and urinary disorders) | 4 (4)
Bladder spasms after 24 hours (Renal and urinary disorders) | 1 (1)
Urethral discomfort after 24 hours (Renal and urinary disorders) | 1 (1)
Pelvic tenderness after 24 hours (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No